CLINICAL TRIAL: NCT06505967
Title: Effectiveness of Qualia NAD+ Supplementation on Intracellular NAD Levels: A Randomized Double-Blind Parallel Trial
Brief Title: Effectiveness of Qualia NAD+ Supplementation on Intracellular NAD Levels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qualia Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NHC-004
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: NAD+ Levels in the Blood

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qualia NAD+ (Experimental)
  Interventions: Dietary Supplement: Qualia NAD+
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Qualia NAD+ — Qualia NAD+ is a novel dietary supplement, formulated to support the maintenance and enhancement of intracellular NAD levels.
  Arms: Qualia NAD+
Other: Placebo — Rice flour
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine if Qualia NAD+ effectively increases NAD+ levels in the blood and to evaluate its safety.

Researchers will compare Qualia NAD+ to a placebo (a look-alike substance that contains no active drug) to assess its efficacy in increasing NAD+ levels in the blood.

Participants will:

Take Qualia NAD+ or a placebo every day for 4 weeks. Undergo blood tests before and after the trial.

ELIGIBILITY:
Inclusion criteria:

Provide voluntary, written, informed consent to participate in the study Agree to provide a valid cell phone number and are willing to receive communications through text.

Healthy male and female participants between the ages of 40-65 years of age. Willingness to complete questionnaires, records, and diaries associated with the study.

Willing to not consume any supplements, energy drinks/shots, or other products containing any form of supplemental vitamin B3 (e.g., niacin, niacinamide, nicotinamide ribosome, NMN) starting about 2 weeks prior to the baseline NAD fingerstick test and continuing through the intervention period.

Willing to not begin taking any new supplements during the study period, and to continue taking any supplements they are currently using regularly (with the exception of vitamin B3 containing supplements).

Willingness to self-administer the intracellular NAD fingerstick test kit at home for both a baseline and post-intervention blood sample, and to complete a release form that gives researchers access to the results of these tests.

Exclusion criteria:

Women who are pregnant, breastfeeding, or planning to become pregnant during the trial Known food intolerances/allergy to any ingredients in the product Having any of the following conditions: Psychiatric conditions, neurologic disorders, endocrine disorders, cancer Having had a significant cardiovascular event in the past 6 months Taking MAO inhibitors, SSRIs, or any other psychiatric or neurological medicines On immunosuppressive therapy Individuals who were deemed incompatible with the test protocol Adults lacking capacity to consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-08-18 (Estimated); Study Completion 2024-09-09 (Estimated)

PRIMARY OUTCOMES:
NAD+ Levels in the Blood | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Qualia Life Sciences, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared